CLINICAL TRIAL: NCT02698956
Title: Edwards SAPIEN 3 Aortic Bioprosthesis Multi-Region Outcome Registry
Brief Title: SOURCE 3: Observational Study to Evaluate Safety and Performance of SAPIEN 3 THV System in Real Life Practice
Acronym: SOURCE 3
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-01
Record Dates: First submitted 2015-02-27; First posted 2016-03-04 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Aortic Stenosis
Keywords: SAPIEN 3 THV; TAVI; Transfemoral; Transaortic; Transapical; Aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TAVI (Transcatheter Aortic Valve Implantation) — Edwards SAPIEN 3 Transcatheter Heart Valve (S3 THV) and Edwards Commander Delivery system (transfemoral) and Certitude Delivery system (transapical/transaortic). The Edwards S3 THV is indicated for use in patients with severe, symptomatic, calcific aortic stenosis with STS Score ≥ 8 or Logistic EuroSCORE ≥15
  Other Names: TAVR

SUMMARY:
This is an international, mutli-center, prospective, consecutively enrolled, observational registry. 2000 patients are planned to be enrolled over one year at up to 150 participating sites.

300 patients out of the 2000 patients enrolled in the main registry are planned to be consecutively enrolled in a select few sites for studying the valve performance. Echocardiogram and angiogram will be taken routinely.

DETAILED DESCRIPTION:
The purpose of this registry is to provide clinical outcome and safety information on patients that will be treated with the Edwards SAPIEN 3 Transcatheter Heart Valve and delivery devices for severe, symptomatic calcific aortic stenosis. In addition, the information collected will serve post market safety and surveillance regulatory obligations.

Consecutive patient data will be collected at baseline, procedure, discharge, after discharge (at approx. 30 days post-index procedure), 12 months post-index procedure and annually thereafter up to 5 years post-implant according to usual practice at site.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from severe, symptomatic, calcific aortic stenosis
* STS Score ≥ 8
* Logistic EuroSCORE ≥15

Exclusion Criteria:

* Congenital unicuspid or congenital bicuspid aortic valve
* Evidence of intracardiac mass, thrombus or vegetation
* Active infection or endocarditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from severe aortic stenosis. Inclusion criteria are based on the decision of the Heart Team.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Olaf Wendler, MD, Principal Investigator — King's College Hospital NHS Trust; Prof. Dr. Alec Vahanian, MD, Principal Investigator — Bichat Hospital
Locations (73):
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
- France (28):
  - CHU Angers, Angers
  - Hopital Jean Minjoz - Besancon, Besançon
  - Clinique Saint-Augustin - Bordeaux, Bordeaux
  - CHU La Cavalle Blanche - Brest, Brest
  - CHU Gabriel-Montpied - Clermont Ferrand, Clermont-Ferrand
  - CHU Bocage - Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hopital Prive Parly II - Le Chesnay, Le Chesnay
  - Centre Chirurgical Marie Lannelongue - Le Plessis-Robinson, Le Plessis-Robinson
  - CHRU Lille, Lille
  - Polyclinique Bois - Lille, Lille
  - Hospices Civiles de Lyon, Lyon
  - Hospices Civils de Lyon, Lyon
  - CHU La Timone - Marseille, Marseille
  - Clinique Clairval - Marseille, Marseille
  - Hopital Saint Joseph - Marseille, Marseille
  - Institut Hospitalier Jacques Cartier Massy, Massy
  - C.H.U. de Nancy, Nancy
  - Clinique Ambroise Pare - Neuilly, Neuilly-sur-Seine
  - CH Pitie Salpetriere, Paris
  - Institut Mutualiste Montsouris - Paris, Paris
  - Hopital Bichat Paris, Paris
  - CHU Hopital Charles Nicolle Rouen, Rouen
  - Centre Cardiologique du Nord - Saint-Denis, Saint-Denis
  - CHU Nantes-Laennec, Saint-Herblain
  - CHRU Strasbourg, Strasbourg
  - CHU Rangueil Toulouse, Toulouse
  - Clinique Saint-Gatien - Tours, Tours
- Germany (26):
  - Klinikum Augsburg, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik GmbH Bad Nauheim, Bad Nauheim
  - Herz und Gefaess Klinik - Bad Neustadt, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Schuechtermann Klinik Bad Rothenfelde, Bad Rothenfelde
  - Herzzentrum Bad Segeberg, Bad Segeberg
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Uniklinik Koeln - Herzzentrum, Cologne
  - Evangelisches Klinikum Niederrhein Herzzentrum Duisburg, Duisburg
  - Universitaetsklinik Erlangen, Erlangen
  - Asklepios Klinik St Georg Hamburg, Hamburg
  - Universitares Herzzentrum Hamburg, Hamburg
  - Klinikum Karlsburg der Klinikgruppe Dr. Guth GmbH & Co. KG, Karlsburg
  - Staedtisches Klinikum Karlsruhe GmbH (SKK), Karlsruhe
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Deutsches Herzzentrum Muenchen (DHM), München
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Regensburg, Regensburg
  - Helios Klinikum Siegburg, Siegburg
  - Robert-Bosch Hospital Stuttgart, Stuttgart
  - Universitaetsklinikum Ulm, Ulm
- Italy (3):
  - Ospedale San Raffaele Milano, Milan
  - Centro Cardiologico Monzino Milano, Milan
  - Azienda A.R.N.A.S. Ospedale Civico di Palermo, Palermo
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Narodny ustav srdcovych a cievnych chorob, a. s., Bratislava, Slovakia
- Policlinica Gipuzkoa Hospital, San Sebastián, Spain
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Klinik im Park Zuerich, Zurich
  - HerzKlinik Hirslanden HKH - Zuerich, Zurich
- United Kingdom (6):
  - Queen Elisabeth Hospital Birmingham, Birmingham
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - St. Thomas Hospital London, London
  - King´s College Hospital London, London
  - Derriford Hospital Plymouth, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarantini G, Nai Fovino L, Le Prince P, Darremont O, Urena M, Bartorelli AL, Vincent F, Hovorka T, Alcala Navarro Y, Dumonteil N, Ohlmann P, Wendler O. Coronary Access and Percutaneous Coronary Intervention Up to 3 Years After Transcatheter Aortic Valve Implantation With a Balloon-Expandable Valve. Circ Cardiovasc Interv. 2020 Jul;13(7):e008972. doi: 10.1161/CIRCINTERVENTIONS.120.008972. Epub 2020 Jun 25. PMID 32580586
- [Derived] Fernandez-Santos S, Theron A, Pibarot P, Collart F, Gilard M, Urena M, Hovorka T, Kahlert P, Zamorano Gomez JL. Valve hemodynamic performance and myocardial strain after implantation of a third-generation, balloon-expandable, transcatheter aortic valve. Cardiol J. 2020;27(6):789-796. doi: 10.5603/CJ.a2019.0049. Epub 2019 May 20. PMID 31106841
- [Derived] Tarantini G, Lefevre T, Terkelsen CJ, Frerker C, Ohlmann P, Mojoli M, Eltchaninoff H, Pinaud F, Redwood S, Windecker S. One-Year Outcomes of a European Transcatheter Aortic Valve Implantation Cohort According to Surgical Risk. Circ Cardiovasc Interv. 2019 Jan;12(1):e006724. doi: 10.1161/CIRCINTERVENTIONS.118.006724. PMID 30630356
- [Derived] Frank D, Abdel-Wahab M, Gilard M, Digne F, Souteyrand G, Caussin C, Collart F, Letocart V, Wohrle J, Kuhn C, Hovorka T, Baumgartner H. Characteristics and outcomes of patients </= 75 years who underwent transcatheter aortic valve implantation: insights from the SOURCE 3 Registry. Clin Res Cardiol. 2019 Jul;108(7):763-771. doi: 10.1007/s00392-018-1404-2. Epub 2018 Dec 14. PMID 30552511
- [Derived] Wendler O, Schymik G, Treede H, Baumgartner H, Dumonteil N, Neumann FJ, Tarantini G, Zamorano JL, Vahanian A. SOURCE 3: 1-year outcomes post-transcatheter aortic valve implantation using the latest generation of the balloon-expandable transcatheter heart valve. Eur Heart J. 2017 Sep 21;38(36):2717-2726. doi: 10.1093/eurheartj/ehx294. PMID 28605423